CLINICAL TRIAL: NCT06483789
Title: Efficacy and Safety of HB-1 for Panic Disorder: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of HB-1 for Panic Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Honeybrains Biotech LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HB-PD-002
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Panic Disorder; Mental Illness
MeSH Terms: conditions — Panic Disorder; Mental Disorders | interventions — Telmisartan; Verapamil; Dosage Forms

STUDY DESIGN:
Intervention Model Description: A sample size of 240 patients (up to a maximum of 600) is planned for the study to be randomized in a 3:1:1:1 ratio of active to monotherapy to monotherapy to placebo control.
Who Masked: Participant, Care Provider, Investigator
Masking Description: An unblinded pharmacist will be utilized to assign bottles to each patient using an interactive voice response system (IVRS) central randomization system. Study treatment or placebo will be dispensed to patients in blinded bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- HB-1 (Experimental): HB-1 fixed dose, once daily.
  Interventions: Drug: HB-1
- Telmisartan (Experimental): Telmisartan fixed dose, once daily.
  Interventions: Drug: Telmisartan Only Product in Oral Dose Form
- Verapamil (Experimental): Verapamil fixed dose, once daily.
  Interventions: Drug: Verapamil Only Product in Oral Dose Form
- Placebo (Placebo Comparator): Placebo treatment, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HB-1 — HB-1 will be supplied as a dual active pharmaceutical ingredient tablet.
  Other Names: Fixed dose Telmisartan / Verapamil tablet
  Arms: HB-1
Drug: Telmisartan Only Product in Oral Dose Form — Telmisartan will be supplied as a single active pharmaceutical ingredient tablet.
  Other Names: Telmisartan
  Arms: Telmisartan
Drug: Verapamil Only Product in Oral Dose Form — Verapamil will be supplied as a single active pharmaceutical ingredient tablet.
  Other Names: Verapamil
  Arms: Verapamil
Drug: Placebo — Matched Placebo will be supplied as a tablet.
  Other Names: Matched Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of HB-1, versus placebo and two monotherapies, in male and female adult patients aged 18 to 65 years, inclusive, with Panic Disorder.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial. All patients with Panic Disorder, with or without specified co-morbidities, who meet all of the inclusion and none of the exclusion criteria will be eligible. Patients and researchers will be blinded to their treatment group.

The study will enroll approximately 240 (up to 600) adult patients who meet the diagnosis of panic disorder.

Patients will be treated for 12 weeks followed by a safety follow up visit one week after their last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 years old, inclusive, at the time of informed consent.
2. Meets Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) Criteria for Panic Disorder.
3. Minimum of one full, unexpected panic attack in week prior to screening (via Diagnostic and Statistical Manual of Mental Disorders 5th edition [DSM-V] based structured interview).
4. Medically stable on current medication regimen for at least 3 months (including as needed [PRN] medications), as determined by Investigator.
5. Willing to remain on current doses of other psychiatric medications throughout the length of the trial.
6. Willing and able to safely stop / avoid any of the following prior to study trial: Inhibitors or inducers of CYP3A4 (grapefruit juice, erythromycin, ritonavir, telithromycin, rifampin), HMG-CoA Reductase Inhibitors (Simvastatin, Lovastatin, Atorvastatin), Beta Blockers (Timolol eyedrops, Metoprolol), Neuromuscular Blocking Agents (curare-like and depolarizing), Antihypertensive Agents (Prazosin and vasodilators, angiotensin-converting enzyme inhibitors, diuretics, beta blockers), Inhalation Anesthetics, Disopyramide, Flecainide, Quinidine, Cimetidine, Lithium, Carbamazepine, Phenobarbital, Cyclosporine, Digitalis, Aliskiren, Ramipril and Ramiprilat, aspirin, propranolol.
7. Willing and able to safely stop / avoid sensitive P-glycoprotein inhibitors.
8. Willing to take HB-1, telmisartan, verapamil, or placebo.
9. Willing and able to provide informed consent indicating an understanding of the requirements of the study and a willingness to comply with scheduled visits and all study procedures.
10. Female subjects must be surgically sterile (or have a monogamous partner who is surgically sterile) or be at least 2 years postmenopausal or commit to use 2 acceptable forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 4 months following the last dose of study treatment. Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms ± spermicide) for the duration of the study and for 4 months following the last dose of study treatment. Individuals who are involved exclusively in same-sex relationships are exempt from the birth control requirements but must agree to abide by the recommendations if they do engage in a heterosexual relationship.
11. Female subjects who are women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening, within 7 days of dosing with study treatment.

Exclusion Criteria:

1. Any concomitant disease, condition, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the participant in the study or interfere with the interpretation of study data.
2. Concurrent treatment with benzodiazepines (e.g. alprazolam, diazepam, clonazepam, lorazepam) as assessed by clinical interview and urine toxicology testing.
3. Severe Agoraphobia (Panic Disorder Symptom Severity Scale (PDSS) Item 4 "agoraphobic fear/avoidance" > 2).
4. Severe Generalized Anxiety (Hamilton Anxiety Rating Scale [HAM-A] Total Score > 23).
5. Prior lifetime history of suicide attempt, Columbia Suicide Severity Rating Scale (C-SSRS) ≥ 4 in the past 6 months or prior lifetime history of hospitalization for depression.
6. Diagnosis of Substance Use Disorder, Obsessive-Compulsive Disorder (OCD), Bipolar I, Bipolar II disorder or schizoaffective or other psychotic disorders (per Structure Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) [SCID-V].
7. Severe uncontrolled cardiac disease within 6 months of Screening, including but not limited to uncontrolled hypertension, hypotension (defined as below 90/60); unstable angina; myocardial infarction (MI) or cerebrovascular accident (CVA).
8. Any clinically significant electrocardiogram (ECG) abnormalities at screening.
9. Inadequate hepatic function defined as total bilirubin > 1.5 × the upper limit of normal (ULN) ranges of each institution, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 3 × the ULN range of each institution.
10. Inadequate renal function defined as serum creatinine > 1.5 × the upper limit of normal (ULN) range of each institution and/or estimated glomerular filtration rate (eGFR) < 60.
11. Any clinically significant abnormalities in clinical laboratory assessments as assessed by the Investigator.
12. Any other systemic conditions or organ abnormalities that in the opinion of the Investigator may interfere with the conduct and/or interpretation of the current study.
13. Unable to complete neuropsychological testing.
14. Already on treatment with either telmisartan or verapamil or both.
15. Has a history of hypersensitivity or severe allergic reaction to either telmisartan or verapamil, or any component of either licensed drug.
16. Documented contraindication to taking telmisartan or verapamil: (e.g., Duchenne's muscular dystrophy, myasthenia gravis).
17. Pregnant or breastfeeding.
18. Participation in another current clinical trial or prior trial within the last three months.
19. Urinalysis evidence of exposure to substances that may interfere with HB-1 testing (per investigator discretion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Unexpected Panic Attacks | Screening, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, and Week 12
  Efficacy will be evaluated through a comparison of the number of unexpected panic attacks from Screening as compared to protocol-specified timepoints per protocol.
Incidence of Treatment-Emergent Adverse Events | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12 and Week 13.
  Safety will be evaluated through the monitoring of Adverse Events and the review of clinically significant changes in routine laboratory tests, ECGs, and orthostatic vital signs.

SECONDARY OUTCOMES:
Change in Clinical Global Impression-Severity Scale (CGI-S) | Baseline, Week 4, Week 8 and Week 12
  Efficacy will be evaluated through an evaluation in Clinical Global Impression Severity scale (CGI-S) scores from Baseline as compared to protocol-specified timepoints per protocol. The Clinical Global Impression Severity Scale is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).
Change in Panic Disorder Symptom Severity Scale (PDSS) | Screening, Week 4, Week 8 and Week 12
  Efficacy will be evaluated through an evaluation in Panic Disorder Symptom Severity Scale (PDSS) scores from Screening as compared to protocol-specified timepoints per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Malcolm Hopwood, Principal Investigator — Ramsay Clinic Albert Road
Locations (22):
- Australia (22):
  - Paratus Clinical Research Canberra, Canberra, Australian Capital Territory
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Novatrials, Kotara, New South Wales
  - Canopy Clinical Sutherland, Miranda, New South Wales
  - Innovate Clinical Research, Waitara, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Canopy Clinical Wollongong, Wollongong, New South Wales
  - Paratus Clinical Research Brisbane, Herston, Queensland
  - Mackay Hospital and Health Service, Mackay, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - South Australian Health and Medical Research Institute, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Grampians Health, Ballarat, Victoria
  - NeuroCentrix, Carlton, Victoria
  - Peninsula Therapeutic and Research Group, Frankston, Victoria
  - Multidisciplinary Alfred Psychiatry Research Clinic, Melbourne, Victoria
  - Ramsay Clinic Albert Road, Melbourne, Victoria
  - Paratus Clinical Research Melbourne, Northcote, Victoria
  - Clinitrials, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No